CLINICAL TRIAL: NCT01420029
Title: Hospital-Based Phthalate Exposure in Very Low Birth Weight Neonates
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: GCO 11-0664; 0285-7451 (Other: CEHC Pilot Projects Fund)
Record Dates: First submitted 2011-08-17; First posted 2011-08-19 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Low Birth Weight Neonates
Keywords: Low birth weight neonates; Neurodevelopmental outcome; Thyroid dysfunction; Extrauterine growth; Plasticizers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine, whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
In this observational pilot project, the investigators plan to document duration and sources of exposure to plasticizers in infants born at birth weights less than 1500 grams. The investigators will examine the association between exposure to plasticizers and outcomes such as performance on a neurological screening tool, extrauterine growth, and thyroid function.

DETAILED DESCRIPTION:
High levels of exposure to certain plasticizers, specifically, phthalates and Bisphenol-A (BPA) have been shown to affect intelligence and behavior in school-age children, as well as to disrupt growth and some endocrine functions. Items used in the care of infants in the Neonatal Intensive Care Unit (NICU) contain phthalates and BPA. Babies admitted for long periods of time to the NICU, could be exposed to high levels of these potentially harmful plastics. In this study, the investigators are interested in documenting duration and sources of exposure to plasticizers during the NICU admission of infants born weighing less than 1500 grams. The investigators will examine the association between NICU exposure to plasticizers and performance on a neurological screening test that predicts future behavior, growth after birth, and the presence of any thyroid dysfunction.

The investigators plan to enroll 50 neonates in our study. The investigators will catalog all exposure to plasticizers during the infant's NICU admission and assign each baby a risk level of exposure. The investigators will then test each infant's performance on a neurological screening tool, measure growth from birth and assess whether or not each infant has thyroid dysfunction and correlate each outcome with exposure risk level. The investigators will also collect urine samples from each baby to store for possible future analysis.

The investigators hypothesize that neonates with higher levels of exposure will demonstrate worse performance on the neurological screening tool, poor growth, and abnormal thyroid function.

ELIGIBILITY:
Inclusion Criteria:

* Neonates born less than 1500 grams that are admitted to the Mount Sinai Hospital NICU

Exclusion Criteria:

* Chromosomal abnormality or other genetic disorder
* Diagnosis of hypoxic-ischemic encephalopathy
* Inborn error of metabolism
* Congenital renal disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Neonates born at birthweights less than 1500 grams will be included.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2011-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Exposure to plasticizers | Length of stay in NICU which averages 8-10 weeks
  Extent of exposure to plasticizers
Performance on neonatal neurological screening tool | 4 weeks of age
Performance on neonatal neurological screening tool | 34 weeks postconceptual age

SECONDARY OUTCOMES:
Extrauterine growth | Weekly during NICU stay with average stay of 8-10 weeks
  Weight, head circumference and length will be recorded weekly during the neonate's stay in the NICU
Thyroid dysfunction | 4 weeks of age
  Presence of thyroid dysfunction on thyroid function tests

CONTACTS AND LOCATIONS:
Overall Officials: Annemarie Stroustrup, MD, MPH, Principal Investigator — Mount Sinai Hospital Division of Newborn Medicine
Locations (1):
- Mount Sinai Hospital Neonatal Intensive Care Unit, New York, New York, United States

REFERENCES:
- [Background] Cho SC, Bhang SY, Hong YC, Shin MS, Kim BN, Kim JW, Yoo HJ, Cho IH, Kim HW. Relationship between environmental phthalate exposure and the intelligence of school-age children. Environ Health Perspect. 2010 Jul;118(7):1027-32. doi: 10.1289/ehp.0901376. Epub 2010 Mar 1. PMID 20194078
- [Background] Wolff MS, Engel SM, Berkowitz GS, Ye X, Silva MJ, Zhu C, Wetmur J, Calafat AM. Prenatal phenol and phthalate exposures and birth outcomes. Environ Health Perspect. 2008 Aug;116(8):1092-7. doi: 10.1289/ehp.11007. PMID 18709157
- [Background] Engel SM, Miodovnik A, Canfield RL, Zhu C, Silva MJ, Calafat AM, Wolff MS. Prenatal phthalate exposure is associated with childhood behavior and executive functioning. Environ Health Perspect. 2010 Apr;118(4):565-71. doi: 10.1289/ehp.0901470. Epub 2010 Jan 8. PMID 20106747
- [Background] Calafat AM, Needham LL, Silva MJ, Lambert G. Exposure to di-(2-ethylhexyl) phthalate among premature neonates in a neonatal intensive care unit. Pediatrics. 2004 May;113(5):e429-34. doi: 10.1542/peds.113.5.e429. PMID 15121985
- [Background] Calafat AM, Weuve J, Ye X, Jia LT, Hu H, Ringer S, Huttner K, Hauser R. Exposure to bisphenol A and other phenols in neonatal intensive care unit premature infants. Environ Health Perspect. 2009 Apr;117(4):639-44. doi: 10.1289/ehp.0800265. Epub 2008 Dec 10. PMID 19440505
- [Background] Weuve J, Sanchez BN, Calafat AM, Schettler T, Green RA, Hu H, Hauser R. Exposure to phthalates in neonatal intensive care unit infants: urinary concentrations of monoesters and oxidative metabolites. Environ Health Perspect. 2006 Sep;114(9):1424-31. doi: 10.1289/ehp.8926. PMID 16966100
- [Background] Loff S, Kabs F, Witt K, Sartoris J, Mandl B, Niessen KH, Waag KL. Polyvinylchloride infusion lines expose infants to large amounts of toxic plasticizers. J Pediatr Surg. 2000 Dec;35(12):1775-81. doi: 10.1053/jpsu.2000.19249. PMID 11101735
- [Background] Subotic U, Hannmann T, Kiss M, Brade J, Breitkopf K, Loff S. Extraction of the plasticizers diethylhexylphthalate and polyadipate from polyvinylchloride nasogastric tubes through gastric juice and feeding solution. J Pediatr Gastroenterol Nutr. 2007 Jan;44(1):71-6. doi: 10.1097/01.mpg.0000237939.50791.4b. PMID 17204957
- [Background] Kim BN, Cho SC, Kim Y, Shin MS, Yoo HJ, Kim JW, Yang YH, Kim HW, Bhang SY, Hong YC. Phthalates exposure and attention-deficit/hyperactivity disorder in school-age children. Biol Psychiatry. 2009 Nov 15;66(10):958-63. doi: 10.1016/j.biopsych.2009.07.034. Epub 2009 Sep 12. PMID 19748073
- [Background] Johnson S, Hollis C, Kochhar P, Hennessy E, Wolke D, Marlow N. Psychiatric disorders in extremely preterm children: longitudinal finding at age 11 years in the EPICure study. J Am Acad Child Adolesc Psychiatry. 2010 May;49(5):453-63.e1. PMID 20431465
- [Background] Tanaka T. Reproductive and neurobehavioural effects of bis(2-ethylhexyl) phthalate (DEHP) in a cross-mating toxicity study of mice. Food Chem Toxicol. 2005 Apr;43(4):581-9. doi: 10.1016/j.fct.2005.01.001. PMID 15721206
- [Background] Price SC, Chescoe D, Grasso P, Wright M, Hinton RH. Alterations in the thyroids of rats treated for long periods with di-(2-ethylhexyl) phthalate or with hypolipidaemic agents. Toxicol Lett. 1988 Jan;40(1):37-46. doi: 10.1016/0378-4274(88)90181-6. PMID 3341048
- [Background] Sugiyama S, Shimada N, Miyoshi H, Yamauchi K. Detection of thyroid system-disrupting chemicals using in vitro and in vivo screening assays in Xenopus laevis. Toxicol Sci. 2005 Dec;88(2):367-74. doi: 10.1093/toxsci/kfi330. Epub 2005 Sep 22. PMID 16179385
- [Background] Silva MJ, Reidy JA, Herbert AR, Preau JL Jr, Needham LL, Calafat AM. Detection of phthalate metabolites in human amniotic fluid. Bull Environ Contam Toxicol. 2004 Jun;72(6):1226-31. doi: 10.1007/s00128-004-0374-4. No abstract available. PMID 15362453
- [Background] Brazelton T, Nugent J. Neonatal Behavioral Assessment Scale, 3rd edition. 1995. Cambridge: MacKeith Press.
- [Background] Engel SM, Berkowitz GS, Barr DB, Teitelbaum SL, Siskind J, Meisel SJ, Wetmur JG, Wolff MS. Prenatal organophosphate metabolite and organochlorine levels and performance on the Brazelton Neonatal Behavioral Assessment Scale in a multiethnic pregnancy cohort. Am J Epidemiol. 2007 Jun 15;165(12):1397-404. doi: 10.1093/aje/kwm029. Epub 2007 Apr 3. PMID 17406008
- [Background] Engel SM, Zhu C, Berkowitz GS, Calafat AM, Silva MJ, Miodovnik A, Wolff MS. Prenatal phthalate exposure and performance on the Neonatal Behavioral Assessment Scale in a multiethnic birth cohort. Neurotoxicology. 2009 Jul;30(4):522-8. doi: 10.1016/j.neuro.2009.04.001. Epub 2009 Apr 16. PMID 19375452
- [Background] Fenster L, Eskenazi B, Anderson M, Bradman A, Hubbard A, Barr DB. In utero exposure to DDT and performance on the Brazelton neonatal behavioral assessment scale. Neurotoxicology. 2007 May;28(3):471-7. doi: 10.1016/j.neuro.2006.12.009. Epub 2007 Jan 10. PMID 17287022
- [Background] Ohgi S, Arisawa K, Takahashi T, Kusumoto T, Goto Y, Akiyama T, Saito H. Neonatal behavioral assessment scale as a predictor of later developmental disabilities of low birth-weight and/or premature infants. Brain Dev. 2003 Aug;25(5):313-21. doi: 10.1016/s0387-7604(02)00233-4. PMID 12850509
- [Background] Clark RH, Thomas P, Peabody J. Extrauterine growth restriction remains a serious problem in prematurely born neonates. Pediatrics. 2003 May;111(5 Pt 1):986-90. doi: 10.1542/peds.111.5.986. PMID 12728076
- [Background] Tamaru S, Kikuchi A, Takagi K, Wakamatsu M, Ono K, Horikoshi T, Kihara H, Nakamura T. Neurodevelopmental outcomes of very low birth weight and extremely low birth weight infants at 18 months of corrected age associated with prenatal risk factors. Early Hum Dev. 2011 Jan;87(1):55-9. doi: 10.1016/j.earlhumdev.2010.10.004. PMID 21078549
- [Background] De Curtis M, Rigo J. Extrauterine growth restriction in very-low-birthweight infants. Acta Paediatr. 2004 Dec;93(12):1563-8. doi: 10.1080/08035250410022198. PMID 15841762
- [Background] Ferguson SA, Flynn KM, Delclos KB, Newbold RR. Maternal and offspring toxicity but few sexually dimorphic behavioral alterations result from nonylphenol exposure. Neurotoxicol Teratol. 2000 Jul-Aug;22(4):583-91. doi: 10.1016/s0892-0362(00)00071-4. PMID 10974597
- [Background] Hinton RH, Mitchell FE, Mann A, Chescoe D, Price SC, Nunn A, Grasso P, Bridges JW. Effects of phthalic acid esters on the liver and thyroid. Environ Health Perspect. 1986 Dec;70:195-210. doi: 10.1289/ehp.8670195. PMID 3830106
- [Background] Pereira C, Mapuskar K, Vaman Rao C. A two-generation chronic mixture toxicity study of Clophen A60 and diethyl phthalate on histology of adrenal cortex and thyroid of rats. Acta Histochem. 2007;109(1):29-36. doi: 10.1016/j.acthis.2006.09.008. Epub 2006 Nov 17. PMID 17113135
- [Derived] Stroustrup A, Bragg JB, Spear EA, Aguiar A, Zimmerman E, Isler JR, Busgang SA, Curtin PC, Gennings C, Andra SS, Arora M. Cohort profile: the Neonatal Intensive Care Unit Hospital Exposures and Long-Term Health (NICU-HEALTH) cohort, a prospective preterm birth cohort in New York City. BMJ Open. 2019 Nov 25;9(11):e032758. doi: 10.1136/bmjopen-2019-032758. PMID 31772104